CLINICAL TRIAL: NCT03536936
Title: Oxygenation and Perfusion in Patients With Acute Migraine Attacks
Acronym: OPAMA
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: Migraine Brain Perfusion
Record Dates: First submitted 2018-05-14; First posted 2018-05-25 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Migraine; Migraine With Aura; Migraine; Status
MeSH Terms: conditions — Migraine Disorders; Migraine with Aura

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to retrospectively evaluate brain perfusion and oxygenation in acute migraine attacks. Magnetic resonance perfusion and susceptibility weighted imaging are the technics to measure perfusion and oxygenation respectively.

DETAILED DESCRIPTION:
The aim of the study is to demonstrate a possible correlation between areas of hypoperfusion and prominent cortical veins during migraine attacks.

These focal ares of altered vascular supply of the brain will be evaluated for correlation with topograhy of symptoms.

ELIGIBILITY:
Inclusion Criteria:

final clinical diagnosis of migraine

Exclusion Criteria:

brain tumors, seizures/epilepsy, confirmed cerebral infarct from cerebral atery occlusion, sinus vein thrombosis;

Ages: 6 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients who present to hospital emergency with acute symptoms of stroke, undergo MR imaging to exclude stroke or other stroke mimics, and at discharge have confirmed diagnosis of acute migraine attack.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Focal cerebral hypoperfusion and elevated oxygenation in acute migraine attack | Patients, who are admitted to hospital, undergo magnetic resonance imaging within 5 days of migraine attack; time frame: symptoms to imaging : 5 days;
  Focal cerebral hypoperfusion and elevated oxygenation in acute migraine attack, measured with visual scores on imaging, using a consensus between two readers

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bosemani T, Burton VJ, Felling RJ, Leigh R, Oakley C, Poretti A, Huisman TA. Pediatric hemiplegic migraine: role of multiple MRI techniques in evaluation of reversible hypoperfusion. Cephalalgia. 2014 Apr;34(4):311-5. doi: 10.1177/0333102413509432. Epub 2013 Oct 18. PMID 24142848
- [Result] Charles A, Brennan KC. The neurobiology of migraine. Handb Clin Neurol. 2010;97:99-108. doi: 10.1016/S0072-9752(10)97007-3. PMID 20816413
- [Result] Fedak EM, Zumberge NA, Heyer GL. The diagnostic role for susceptibility-weighted MRI during sporadic hemiplegic migraine. Cephalalgia. 2013 Nov;33(15):1258-63. doi: 10.1177/0333102413491027. Epub 2013 Jun 13. PMID 23766355
- [Result] Floery D, Vosko MR, Fellner FA, Fellner C, Ginthoer C, Gruber F, Ransmayr G, Doerfler A, Uder M, Bradley WG. Acute-onset migrainous aura mimicking acute stroke: MR perfusion imaging features. AJNR Am J Neuroradiol. 2012 Sep;33(8):1546-52. doi: 10.3174/ajnr.A3020. Epub 2012 Apr 19. PMID 22517281
- [Result] Forster A, Wenz H, Kerl HU, Brockmann MA, Groden C. Perfusion patterns in migraine with aura. Cephalalgia. 2014 Oct;34(11):870-6. doi: 10.1177/0333102414523339. Epub 2014 Feb 19. PMID 24554619
- [Result] Kao HW, Tsai FY, Hasso AN. Predicting stroke evolution: comparison of susceptibility-weighted MR imaging with MR perfusion. Eur Radiol. 2012 Jul;22(7):1397-403. doi: 10.1007/s00330-012-2387-4. Epub 2012 Feb 10. PMID 22322311
- [Result] Launer LJ, Terwindt GM, Ferrari MD. The prevalence and characteristics of migraine in a population-based cohort: the GEM study. Neurology. 1999 Aug 11;53(3):537-42. doi: 10.1212/wnl.53.3.537. PMID 10449117
- [Result] Mourand I, Menjot de Champfleur N, Carra-Dalliere C, Le Bars E, Roubertie A, Bonafe A, Thouvenot E. Perfusion-weighted MR imaging in persistent hemiplegic migraine. Neuroradiology. 2012 Mar;54(3):255-60. doi: 10.1007/s00234-011-0946-z. Epub 2011 Aug 11. PMID 21833737
- [Result] Planche V, Chassin O, Leduc L, Regnier W, Kelly A, Colamarino R. Sturge-Weber syndrome with late onset hemiplegic migraine-like attacks and progressive unilateral cerebral atrophy. Cephalalgia. 2014 Jan;34(1):73-7. doi: 10.1177/0333102413505237. Epub 2013 Sep 17. PMID 24045571